CLINICAL TRIAL: NCT00016952
Title: Phase II Study in Patients With Metastatic Colorectal Carcinoma Previously Treated With Oxaliplatin (OXAL) or a Combination of Irinotecan (CPT-11) and OXAL
Brief Title: Irinotecan or Fluorouracil Plus Leucovorin in Treating Patients With Previously Treated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0048; NCI-2012-02383 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068635 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- irinotecan (Experimental): Prior oxaliplatin-based chemotherapy: Patients receive irinotecan IV over 90 minutes on day 1. Treatment repeats every 3 weeks.
  Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with a confirmed complete response for 2 consecutive courses may discontinue treatment at investigator's discretion.
  Quality of life is assessed at baseline, approximately every 6 weeks during treatment, and then after the last course of treatment.
  Patients are followed every 3 months for 5 years.
  Interventions: Drug: irinotecan hydrochloride
- leucovorin + fluorouracil (Experimental): Prior to irinotecan and oxaliplatin combination chemotherapy: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV continuously on days 1 and 2. Treatment repeats every 2 weeks.
  Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with a confirmed complete response for 2 consecutive courses may discontinue treatment at investigator's discretion.
  Quality of life is assessed at baseline, approximately every 6 weeks during treatment, and then after the last course of treatment.
  Patients are followed every 3 months for 5 years.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium

INTERVENTIONS:
Drug: fluorouracil
  Arms: leucovorin + fluorouracil
Drug: irinotecan hydrochloride
  Arms: irinotecan
Drug: leucovorin calcium
  Arms: leucovorin + fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving the drugs in different combinations may kill more tumor cells.

PURPOSE: Phase II trial to compare the effectiveness of either irinotecan or fluorouracil plus leucovorin in treating patients who have metastatic colorectal cancer that has been previously treated with oxaliplatin with or without irinotecan.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the tumor response rate in patients receiving irinotecan or fluorouracil and leucovorin calcium for metastatic colorectal cancer previously treated with oxaliplatin with or without irinotecan.
* Determine the time to tumor progression, time to treatment failure, and overall survival of patients treated with these regimens.
* Determine the toxic effects of these regimens in these patients.
* Evaluate the quality of life of patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy (oxaliplatin-based therapy vs irinotecan and oxaliplatin combination therapy). Patients are assigned to one of two treatment groups.

* Group I (prior oxaliplatin-based chemotherapy): Patients receive irinotecan IV over 90 minutes on day 1. Treatment repeats every 3 weeks.
* Group II (prior irinotecan and oxaliplatin combination chemotherapy): Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV continuously on days 1 and 2. Treatment repeats every 2 weeks.
* Both groups: Treatment continues in the absence of disease progression or unacceptable toxicity. Patients with a confirmed complete response for 2 consecutive courses may discontinue treatment at investigator's discretion.

Quality of life is assessed at baseline, approximately every 6 weeks during treatment, and then after the last course of treatment.

Patients are followed every 3 months for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic colorectal adenocarcinoma incurable by surgery or not amenable to radiotherapy with curative intent
* Progressive disease after one of the following prior treatments for metastatic disease:

  * Oxaliplatin-based chemotherapy
  * Irinotecan and oxaliplatin combination chemotherapy
* At least 1 measurable lesion

  * At least 20 mm in at least one dimension
* No known CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 0.5 mg/dL above upper limit of normal (ULN)
* AST no greater than 5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No unstable angina
* No symptomatic congestive heart failure
* No serious uncontrolled cardiac arrhythmia

Other:

* No active or uncontrolled infection
* No evidence of other serious illness
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or noninvasive carcinomas
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent sargramostim (GM-CSF)

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No more than 1 prior chemotherapy regimen for advanced colorectal cancer
* Prior adjuvant chemotherapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to more than 25% of bone marrow

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-04; Primary Completion 2004-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
tumor response rate | Up to 5 years

SECONDARY OUTCOMES:
time to tumor progression | Up to 5 years
time to treatment failure | Up to 5 years
overall survival | Up to 5 years
quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry C. Pitot, MD, Study Chair — Mayo Clinic
Locations (15):
- United States (14):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada